CLINICAL TRIAL: NCT06952569
Title: Age-Gate Validation Functionality Testing of the IKE Application
Brief Title: Human Factors Validation and Usability Testing of the IKE Age-Gating System
Status: Completed | Type: Observational
Sponsor: IKE Tech (Industry)
Responsible Party: Sponsor
Organization: Ispire Technology, Inc. (Industry)
Other Study IDs: Pro00083344
Record Dates: First submitted 2025-04-18; First posted 2025-05-01 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Vaping; Underage
Keywords: Youth; ENDs; e-cigarette; e-cigarettes; age-gate; age-verify; Bluetooth; BLE; validation; software; IKE; Ispire; Access
MeSH Terms: conditions — Vaping

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (6):
- Age 18-20, non user
  Interventions: Other: IKE System
- Age 21-24, Smoker, Vape user or Both
  Interventions: Other: IKE System
- Age 22-44, Smoker, Vape user or Both
  Interventions: Other: IKE System
- Age 45-64, Smoker, Vape user or Both
  Interventions: Other: IKE System
- Age 65 or older, Smoker, Vape user or Both
  Interventions: Other: IKE System
- Age 65 or older, Non-user
  Interventions: Other: IKE System

INTERVENTIONS:
Other: IKE System — Age-gate the access and activation of a device to authorized users of legal age
  Other Names: IKE Application; IKE Bluetooth; IKE BLE

SUMMARY:
A multi-center human factors validation study to demonstrate the function of the IKE Bluetooth system on a chip (SoC) and mobile applications ability to age-gate a device, accurately identify an individuals age, race/ethnicity, and gender, and asses the usability of the IKE System.

DETAILED DESCRIPTION:
Study Objectives:

IKE developed a smartphone application which identifies and age-verifies users and works in conjunction with a Bluetooth low energy (BLE) chip to restrict connecting to and activating a device by a users age. The intention is to use this in ENDs devices, and therefore the age limit was set to 21 years. This feature is generally referred to as "age-gating."

The purpose of the study is to:

* Generally establish the ability of individuals to successfully download and use the IKE application
* Confirm the identification and age-verification application works effectively to prevent those under 21 from enabling the IKE application
* Confirm the identification and age-verification application works effectively to allow those 21 years of age or older to enable the IKE application
* Establish that only individual over 21 years of age is able to connect a device to the IKE application via Bluetooth

Upon successful Bluetooth connection to the device via the IKE application:

* Confirm the Maximum Idle Time function works by disconnecting the device and powering the device off within a maximum of 15 minutes
* Confirm the Out of Bluetooth Range function works specific to connection of the Vape device to the smartphone (Vape device will be placed in Faraday bag to force disconnect from smartphone) and the user can re-activate the device
* Confirm users are able to reactivate the same device after either Maximum Idle Time disconnect or Out of Bluetooth Range disconnect

Establish the ability of an identity and age-verified individual to log-in to the application on a secondary device (in this case a tablet) and effectively connect the device using Bluetooth while simultaneously forcing disconnection of the previously connected device

Further, the research is designed to have participants use the smartphone application in as natural as possible setting without direct instruction to simulate a real-world use setting.

ELIGIBILITY:
Inclusion Criteria:

1. Currently live in proximity to one of the four central location sites
2. Ages 18 and older
3. Have a valid driver's license or US government-issued identification with picture
4. Currently use a smartphone with an iOS (Apple) or Android operating system
5. Indicate somewhat (3), very (4), or extremely (5) comfortable using smartphone applications on intake questionnaire
6. Able and willing to comply with all study requirements
7. Review and sign informed consent

Exclusion Criteria:

1. Under 18 years of age
2. Among 21-64 years of age, do not currently use cigarettes or vape products
3. Do not own or use a smartphone with an iOS (Apple) or Android operating system
4. Unable to download any smartphone application
5. Employees of or household member employed in advertising/marketing, market research, healthcare, legal field, news and media, or local, state or US Federal government to minimize bias and to protect any proprietary product information that will be disclosed in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: General population
Sampling Method: Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2025-02-18 (Actual); Primary Completion 2025-03-30 (Actual); Study Completion 2025-03-30 (Actual)

PRIMARY OUTCOMES:
Accurately age-verify users using a government ID and live photo | Day 1
  Error rate
Prevents users under 21 year of age from enabling IKE application | Day 1
  Pass or Fail
Allows users age 21 and older to enable IKE application | Day 1
  Pass or Fail
IKE application connects to and activates a device for users over 21 years of age | Day 1
  Pass or Fail
Users are able to download the IKE application | Day 1
  Task completion Error rate
Device disconnects and powers off within 15 minutes of idling (no use) | Day 1
  Pass or Fail
Device is disconnected and powered off after losing Bluetooth signal | Day 1
  Pass or Fail
User is able to reactivate the device after being disconnected and powered off | Day 1
  Task completion

SECONDARY OUTCOMES:
User download the IKE application on personal smartphone | Day 1
  Error rate
Perceived Ease of IKE Application Account Setup | Day 1
  Extremely Easy (1), Very Easy (2), Somewhat Easy (3), Not very easy (4), Not at all easy (5)
Accurately identifies age, race/ethnicity, and gender | Day 1
  Error rate

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Alder Weiner, MARC Research facility partner, Los Angeles, California
  - Focus Center, MARC Research facility partner, Chicago, Illinois
  - L&E Research, MARC Research facility partner, New York, New York
  - Creative Consumer Research, MARC Research facility partner, Houston, Texas

IPD SHARING:
Plan to Share IPD: No